CLINICAL TRIAL: NCT04729231
Title: A Randomized Controlled Trial Comparing the Functional and Aesthetic Outcomes of Lobed Transposition Flaps vs. Nasalis Sling Flaps in Nasal Tip Reconstruction
Brief Title: Reconstruction Flaps for Nasal Surgical Wounds RCT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed before enrollment could begin.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STU00211248
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Surgical Wound
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nasalis Sling Flap (Active Comparator)
  Interventions: Procedure: Nasalis Sling Flap
- Lobed transposition flap (Active Comparator)
  Interventions: Procedure: Lobed Transposition Flap

INTERVENTIONS:
Procedure: Nasalis Sling Flap — The nasalis sling flap involves alteration of the nasalis muscle to create a myocutaneous pedicle flap that will be used to fill in the wound.
  Arms: Nasalis Sling Flap
Procedure: Lobed Transposition Flap — Lobed flap reconstruction involves the use of cutaneous tissue located adjacent to the nasal tip to fill in the wound. The flap will undergo a 90-degree arc to approximate the desired position.
  Arms: Lobed transposition flap

SUMMARY:
The purpose of this study is to determine whether there is a significant difference in aesthetic and functional outcomes between nasalis sling flaps and lobed flaps of nasal tip wounds requiring reconstruction.

This is a randomized clinical trial. Approximately 32 participants who are undergoing nasal tip wound reconstruction surgery will be invited to participate and randomized to receive either the nasalis sling repair or the lobed flap repair. Patients will be asked to complete a few questionnaires including a VAS scale, the Surgical Outcomes scale, the NOSE instrument, and the Nasal Appearance and Function Evaluation Questionnaire (NAFEQ).

This study was a pilot study designed to determine the feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years
* Defect located on the nasal tip, infratip, or supratip of the nose
* Longest length of the wound should be no greater than 15mm
* Participants must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Active infection
* Age <18
* Investigator judgement that patient is not suitable for randomization (preexisting scars or architecture that would make one repair option less likely to be successful)
* Current cigarette smoking
* Patients that have a disease or are taking medication that would severely impair wound healing in the opinion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 6-16 weeks after the procedure
  This visual analog scale (VAS) measures outcomes of functionality and appearance with values ranging on a continuum from 0 to 10, and higher scores representing a better outcome.
Surgical Outcome Scale | 6-16 weeks after the procedure
  The Surgical Outcome Scale is a likert agreement scale on surgical outcomes with values ranging from 1 (agree) to 5 (disagree), and lower scores representing a better outcome.
Nasal Obstruction Symptom Evaluation (NOSE) Instrument | Baseline to 6-16 weeks
  The Nasal Obstruction Symptom Evaluation (NOSE) Instrument is a questionnaire of nose functionality. This is a checklist of of problems related to the nose/nasal area with possible answers ranging from "not a problem" to a "severe problem".
Nasal Appearance and Function Evaluation Questionnaire (NAFEQ) Scale | Baseline to 6-16 weeks
  Nasal Appearance and Function Evaluation Questionnaire (NAFEQ) Scale is a likert scale on nasal appearance and function evaluations with values ranging from 1 (always; very poor; very dissatisfied) to 5 (never; excellent; very satisfied), and higher scores representing a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided